CLINICAL TRIAL: NCT07392359
Title: Prospective, Multicentre, Randomised Controlled, Non-Inferiority Clinical Trial Evaluating the Safety and Efficacy of the TAVR Assist System and Its Disposable Kit for Use as an Adjunct to TAVR
Brief Title: Zhicheng TAVR Robot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhicheng Medical Technology (Jiaxing) Co, Ltd (Industry)
Collaborators: Xiamen Cardiovascular Hospital, Xiamen University (Other); Fu Wai Hospital, Beijing, China (Other); Beijing Anzhen Hospital (Other); The General Hospital of Northern Theater Command (Other); Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1RAD0008
Record Dates: First submitted 2025-11-13; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Aortic Stenosis Treated With TAVI
Keywords: TAVR Assist System; Aortic stenosis treated with TAVI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVR with TAVR Assistance System (Experimental)
  Interventions: Device: TAVR Assistance System
- TAVR By Manual (Placebo Comparator)
  Interventions: Other: TAVR by manual

INTERVENTIONS:
Device: TAVR Assistance System — Whether or not TAVR procedures are performed with a TAVR assist system
  Arms: TAVR with TAVR Assistance System
Other: TAVR by manual — TAVR by manual
  Arms: TAVR By Manual

SUMMARY:
Use of the Transcatheter Aortic Valve Replacement Surgical Assist System and its Disposable Kit in Patients With Severe Aortic Stenosis to Evaluate the Safety and Efficacy of the Transcatheter Aortic Valve Replacement Surgical Assist System and its Disposable Kit for Use as an Adjunct to Transcatheter Aortic Valve Replacement

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old, gender is not limited;
* Patients assessed by a cardiac multidisciplinary team (MDT) expert panel as having severe aortic stenosis and suitable for transcatheter aortic valve replacement;

  *Severe aortic stenosis was defined as echocardiographically demonstrated transaortic valve flow velocity ≥4.0 m/s, or transaortic valve pressure differential ≥40 mmHg (1 mmHg=0.133 kPa), or aortic orifice area <1.0 cm2, or effective aortic orifice area index <0.6 cm2/m2; for low-pressure-differential-low-flow rate by dopa-phenobutylamine loading test, Doppler ultrasound evaluation or other imaging means of assessment for those judged to have severe aortic stenosis.
* Have a core laboratory assessment that the patient is anatomically suitable for transcatheter aortic valve replacement;
* Patients who understand the purpose of the trial, voluntarily participate in the trial, sign an informed consent form, and are willing to cooperate in the follow-up.

Exclusion Criteria:

* Patients whose access or aortic root anatomical pattern is unsuitable for TAVR treatment;
* Poor peripheral arterial conditions that preclude transfemoral TAVR;
* Aortic annulus horizontal pinch angle ≥65° as measured by preoperative MDCT;
* Patients at high risk of coronary obstruction requiring intraoperative coronary protection measures;
* Patients requiring intraoperative delivery with a grapple assist system;
* Previous implantation of a prosthetic aortic valve (bioprosthetic or mechanical);
* Active stage of infective endocarditis or other active infection;
* Combined mitral, tricuspid or severe macrovascular lesions requiring surgical or interventional intervention;
* Echocardiography suggestive of left ventricular thrombus, intracardiac mass or redundant organisms;
* Diagnosis of hypertrophic cardiomyopathy, restrictive cardiomyopathy, infiltrative cardiomyopathy (e.g. amyloidosis, haemochromatosis, nodular disease, etc.), constrictive pericarditis;
* Severe obstruction of the left ventricular outflow tract without corrective measures;
* Severe pulmonary hypertension (pulmonary artery systolic pressure >70 mmHg measured by ultrasound);
* Severe right heart dysfunction as suggested by a combined clinical and ultrasound assessment;
* Severe left heart systolic insufficiency (left ventricular ejection fraction <30%);
* Cardiogenic shock or haemodynamic instability requiring ventricular assist device therapy within 30 days prior to enrolment;
* End-stage heart failure (ACC/AHA Stage D), or post cardiac transplantation, or awaiting cardiac transplantation;
* Acute myocardial infarction within 30 days prior to enrolment;
* Has had a stroke within 3 months prior to enrolment;
* Stenosis of the common or internal carotid artery or vertebral artery (>70% stenosis) requiring treatment as recommended by the relevant disciplinary consultation;
* Severe cardiac and aortic disease requiring concomitant treatment, including ascending aortic aneurysm (maximum diameter ≥ 50 mm);
* Severe renal insufficiency (estimated glomerular filtration rate <30mL/min/1.73m2);
* Active peptic ulcer or history of upper gastrointestinal bleeding within 3 months prior to enrolment;
* Severe coagulopathy; Patients with known intolerance to anticoagulant, antiplatelet drugs or anaesthetic drugs; Patients who have participated in other drug or medical device clinical trials prior to enrolment that have not met the primary endpoint; Patients who, in the opinion of the investigator, are not suitable for participation in this clinical trial

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Technical Success at exit from OR, hybrid room or cath lab post-index procedure | Immediate after procedure
  Absence of procedural mortality; and Successful access, delivery, and retrieval of transcatheter delivery system; and Deployment and correct positioning of a single intended THV; and Freedom from re-intervention related to the device or access procedure

SECONDARY OUTCOMES:
Device Success | 30 days
  Absence of procedure mortality; and Correct position of a single prosthetic heart valve Intended performance of the prosthetic heart valve (i.e., no prosthesis mismatch and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s; and no moderate or severe prosthetic valve regurgitation) Intended performance of the prosthetic heart valve (i.e., no prosthesis mismatch and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s; and no moderate or severe prosthetic valve regurgitation)
Cardiac function changement | Baseline，30 days
  Cardiac function changement is accessed by NYHA cardiac function classification increases from baseline to 30 days
Prosthetic aortic valve function | 1、immediately after the procedure; 2、3 days; 3、30 days
  Effective orifice area, mean transvalvular pressure difference, degree of regurgitation (mid-valve, peri-valve), degree of stenosis, etc.
Duration of aortic valve replacement | During the procedure
  Time from start of delivery of prosthetic aortic valve by valve delivery system to successful implantation of prosthetic aortic valve
Total exposure of the operator to radiation | During the procedure
  The doctor wears radiation detection equipment and records the total radiation exposure during the surgical procedure
Number of surgical staff | During the procedure
Evaluation of Device Performance with questionnaires | immediately after the procedure
  For test group only，using questionnaires to evaluate Device performance

IPD SHARING:
Plan to Share IPD: No